CLINICAL TRIAL: NCT04320303
Title: CMV Infection and Immune Intervention After Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: CMV Infection and Immune Intervention After Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, President, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016PhB175-01
Record Dates: First submitted 2020-03-23; First posted 2020-03-24 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: CMV Viremia; Transplantation Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adaptive NK cells infusion post transplantation (Experimental): Adaptive donors expanded NK cells infusion at day 20±3d and 27±3d post transplantation
  Interventions: Biological: expanded NK cells

INTERVENTIONS:
Biological: expanded NK cells — Donor derived expanded NK cells were infused to patients at around days 20±3d, and 27±3d post transplantation.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective or even the only way to cure blood malignant diseases. Cytomegalovirus (CMV) infection is a serious early complication of allo-HSCT. Its high incidence and poor prognosis can cause a series of terminal organ diseases such as CMV pneumonia, encephalitis, and enteritis,which seriously affecting the prognosis of patients post allo-HSCT.

Our data show that rapid reconstruction of NK cells after transplantation can reduce the incidence of CMV infection. Patients with a rapid reconstruction of NKG2C after transplantation have a low CMV infection rate, and patients with strong secretion of IFN-gamma of NK after transplantation have low CMV infection.

Our previous research showed that trophoblast cells transfected with IL-21 and 4-1BBL can achieve a large number of clinical-grade expansion of NK cells (mIL-21 / 4-1BBL NK cells), and mIL-21 / 4-1BBL NK cells It is safe to treat patients with minimal residual disease (MRD) positive AML after transplantation, and can induce MRD to turn negative. Previous studies have shown that adoptive infusion of expanded NK cells after haplotype transplantation is safe and can improve the functional reconstruction of NK cells. Therefore, we hypothesized that the infusion of NK cells can improve the antiviral capacity of NK cells, thereby effectively reducing the CMV infection. Incidence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute leukemia (AL) or myelodysplastic syndrome (MDS) or myeloma or lymphoma undergoing haploidentical allogeneic stem cell transplantation
2. No CMV infection by 20 days ± 3 days after transplantation
3. No active acute GVHD by 20 days ± 3 days after transplantation
4. The dose of prednisolone was less than 0.5mg / kg / d within 72 hours before and after infusion of NK cells
5. Prior to transplantation, the CMV IgG of the recipient and donor were positive, and the recipient had a suitable donor to expand NK cells.
6. Patient age 16-65 years
7. Donor age 16-65 years
8. Patient Karnofsky score> 70%
9. Estimated survival> 3 weeks
10. Patient agrees to participate in study

Exclusion Criteria:

1. Participants in any other clinical trials within 1 month before enrollment
2. Active infection
3. HBV or HCV or HIV carriers
4. With moderate to severe renal dysfunction (blood creatinine> 130umol / L) and / or liver dysfunction (total bilirubin> 34umol / L, ALT, AST> 2 times the upper limit of normal) before NK infusion
5. Researchers do not consider it appropriate to participate in this trial.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of CMV infection post transplantation | within 180 days post transplantation
  Whether to reduce the incidence of CMV infection in patients post haploidentical transplantation

SECONDARY OUTCOMES:
Cumulative incidence of refractory CMV infection post transplantation | within 180 days post transplantation
  Whether to reduce the incidence of refractory CMV infection in patients post haploidentical transplantation
Cumulative incidence of CMV disease post transplantation | within 180 days post transplantation
  Whether to reduce the incidence of CMV disease in patients post haploidentical transplantation
Enhanced anti-CMV function of reconstituted NK cells | within 180 days post transplantation
  Whether to enhance the anti-CMV function of reconstituted NK cells
cumulative incidence of TRM | within 180 days post transplantation
  Whether to reduce the incidence of transplantation related mortality in patients post haploidentical transplantation
cumulative incidence of overall survival | within 180 days post transplantation
  Whether to increase the incidence of overall survival in patients post haploidentical transplantation
cumulative incidence of disease free survival | within 180 days post transplantation
  Whether to increase the incidence of disease free survival in patients post haploidentical transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No